CLINICAL TRIAL: NCT04496440
Title: Primary Osteoarthritis Knee - Establishing Its Cause, Pathogenesis and Treatment
Brief Title: An Attempt to Find Out Root Cause of a Pain Producing Knee Disease
Status: Completed | Type: Observational
Sponsor: DR R C Agrawal (Other)
Responsible Party: Sponsor-Investigator, DR R C Agrawal, Senior Surgeon, Knee Pain Clinic
Organization: Knee Pain Clinic (Other)
Other Study IDs: 1001
Record Dates: First submitted 2020-06-28; First posted 2020-08-03 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Knee Osteoarthritis; Arthroplasty; Knee
Keywords: Deficient full flexion; Deficient full extension; Contracture Correction Therapy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trial Group: Contracture correction therapy
  Interventions: Other: Contracture Correction Therapy
- Control Group: No new intervention, patients continued with the previous treatment.

INTERVENTIONS:
Other: Contracture Correction Therapy — Non-drug and non-surgical treatment of contracted knee capsules
  Groups: Trial Group

SUMMARY:
This study was focused on a type of arthritis (knee) in which patients develop pain with disabilities in sitting and walking etc. In advance stage the person is bereft of his/her personal physical activities. The prevalent treatment is temporary and dis-satisfactory. A new treatment was designed and a trial was conducted on 125 patients (100 in the trial group, 25 in the control group) for a duration of six months.

DETAILED DESCRIPTION:
The study was focused on establishing the cause and treatment of a painful knee joint disease (Primary Osteoarthritis Knee = OA Knee). At present the cause and treatment are not known. The study was based on a hypothesis, designing a treatment and testing it through a clinical trial. This established that the deficient full flexion or deficient full extension of knee joints, producing contracture in their capsules was the cause and the correction (Contracture Correction Therapy = CCT) was the cure of the disease. The correction was carried out by passive flexion or passive extension of affected knee through eight body postures designed specifically during the study.

To test the efficacy a multi-centre, multi surgeon six months study on 125 patients was carried out, patients were divided into Trial and Control groups. The effects were measured by primary outcome measure - The Western Ontario and McMaster Universities Arthritis Index (WOMAC) score and other measure EuroQol-Visual Analogue Scales (EQ-VAS) score, DFF*, DFE^ at 0, 6 ,12 and 24 weeks.

The "Intervention" for 1st group was CCT and for the 2nd group was "No intervention".

* Deficient full flexion

^ Deficient full extension

ELIGIBILITY:
Inclusion Criteria:

* Age =>30 years
* Knee pain which appeared without any apparent cause, exacerbated by exertion and subsided by rest.
* Presence of limited morning stiffness
* No history of infection, inflammation or trauma to rule out secondary OA
* Disability in sitting, climbing stairs or walking

Exclusion Criteria:

* Backache
* Leg pain (e.g. sciatica)
* Inability to lie supine (e.g. kyphosis)
* Inability to lie prone (e.g. central obesity)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gwalior a city in India and multiple surrounding towns
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
WOMAC Knee Arthritis score | 6 Months
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) on a five point likert-type scale. Range 0-96, 0=BEST and 96=WORST. To access a change from baseline score at six months.

SECONDARY OUTCOMES:
EuroQol visual analogue scale (EQ-VAS) | 6 Months
  A 20 centimetre vertical visual analogue scale (EQ-VAS), that takes values between 100 (best imaginable health) and 0 (worst imaginable health). To access a change from baseline score at six months.
Deficient Full Flexion (DFF) | 6 Months
  The degree by which flexion is lesser then 145°. Full flexion is measured by Goniometer, expressed in blocks of 5°, such as 140°, 135°, 130° etc. In first case DFF is 145-140 = 5°. Higher degree of DFF denotes higher severity. To access a change from baseline score at six months.
Deficient Full Extension (DFE) | 6 Months
  The degree by which full extension falls short to 0°. When full Range of Motion (ROM) is 0-145° and full extension is 145° the Full extension is should be 0.The DFE are represented by 5°, 10°, 15° etc. Higher degree of DFE denotes higher severity. To access a change from baseline score at six months.

CONTACTS AND LOCATIONS:
Overall Officials: R C Agrawal, MBBS,MS,FICS, Principal Investigator — Knee Pain Clinic
Locations (6):
- India (6):
  - Arogya Sadan Nursing Home, Bhind, Madhya Pradesh
  - Sai Baba Dharmarth Chikitsalaya, Gwalior, Madhya Pradesh
  - Parashar Poly Clinic, Gwalior, Madhya Pradesh
  - Knee Pain Clinic, Gwalior, Madhya Pradesh
  - Lok Hitkari Trust Health Camp, Gwalior, Madhya Pradesh
  - Dr. Shukla Surgery Center, Morena, Madhya Pradesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The WOMAC is a widely used self-administered health status measure used in assessing pain, stiffness, and function in patients with OA of the hip or knee. — https://www.orthopaedicscore.com/scorepages/knee_injury_osteopaedic_outcome_score_womac.html
- See also: EuroQol-visual analogue scales - It measure the health status on 20 cms. vertical scale, 0-100, 100 represent best health. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4287662/